CLINICAL TRIAL: NCT00884234
Title: A Phase 2, Double-Blind, Randomized, Parallel-Group, Controlled, Repeat Dose, Single Center Study to Evaluate the Safety and Efficacy of RT001, a Botulinum Toxin Type A Topical Gel, for the Treatment of Moderate to Severe Lateral Canthal Lines In Adults
Brief Title: Safety and Efficacy Study of RT001 to Treat Moderate to Severe Lateral Canthal Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RT001-CL011LCL
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Lateral Canthal Lines
Keywords: Lateral Canthal Lines; Crow's Feet; Facial Wrinkles; Lateral Canthal Area
MeSH Terms: interventions — RT001

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): RT001 (Botulinum Toxin Type A Topical Gel)
  Interventions: Drug: RT001 (Botulinum Toxin Type A Topical Gel)
- 2 (Placebo Comparator): Vehicle Control
  Interventions: Other: Vehicle Control

INTERVENTIONS:
Other: Vehicle Control — Two sequential doses of Vehicle Control at Baseline (Day 0) and Week 2
  Arms: 2
Drug: RT001 (Botulinum Toxin Type A Topical Gel) — Two sequential doses of RT001 at Baseline (Day 0) and Week 2
  Arms: 1

SUMMARY:
The purpose of this study is to determine the safety and efficacy of 2 sequential doses of RT001 compared to vehicle control following applications at Baseline (Day 0) and Week 2.

DETAILED DESCRIPTION:
This is a double-blind, randomized, parallel-group, controlled, repeat dose, single center study to evaluate the safety and efficacy of repeat application of RT001 in at least 30 subjects with moderate to severe lateral canthal lines. Subjects will be randomized to 1 of 2 treatment groups in a 1:1 ratio (RT001 Dose A or vehicle control).

ELIGIBILITY:
Inclusion Criteria:

1. Female/male ages 30 to 55
2. Bilateral lateral canthal lines rated as moderate or advanced.
3. Willing to refrain from any product that affects skin remodeling or a product that may cause an active dermal response in the treatment area beginning at screening through Week 6.
4. Women of child baring potential must practice and be willing to continue to use an effective method of birth control.

Exclusion Criteria:

1. Muscle weakness or paralysis in the area receiving treatment.
2. Active skin disease or irritation at treatment areas.
3. Undergone any procedures that may affect the lateral canthal region during the past 12 months prior to screening.
4. Previous treatment with botulinum toxin (any serotype) in the head or neck area within 9 months prior to Baseline (Day 0).
5. Use of topical steroid on either of the treatment areas or use of medications that suppress the immune system 30 days prior to screening and continuing through End of Study (Week 6).
6. Any abnormality on the electrocardiogram (ECG) at screening or any history of clinically significant arrhythmia, unstable angina, myocardial infarction or congestive hear failure.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The number of subjects classified as exhibiting improvement via the Investigator Global Assessment from Baseline (Day 0) to End of Study (Week 6). | Baseline (Day 0) and Week 6
Incidence of treatment emergent AEs. | Baseline (Day 0) and Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Bruce, MD, Principal Investigator — The Center for Skin Research
Locations (1):
- Suzanne Bruce & Associates / The Center for Skin Research, Houston, Texas, United States